CLINICAL TRIAL: NCT02222129
Title: A Randomized Controlled Trial for Pain Control in Laparoscopic Urologic Surgery: 0.25% Bupivacaine Versus Long-Acting Liposomal Bupivacaine
Brief Title: Efficacy of Liposomal Bupivacaine Versus 0.25% Bupivacaine for Laparoscopic Urologic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Knight, Richard, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 403263-1; BHS120036 (Other: Local IRB)
Record Dates: First submitted 2014-08-19; First posted 2014-08-21 (Estimated); Results first posted 2015-04-16 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Pain, Postoperative
Keywords: Randomized controlled trial; anesthetics-local; bupivacaine; analgesia; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine (Active Comparator): Surgical site infiltration of 0.25% bupivacaine.
  Interventions: Drug: Bupivacaine
- Liposomal bupivacaine (Experimental): Surgical site infiltration of liposomal bupivacaine.
  Interventions: Drug: liposomal bupivacaine

INTERVENTIONS:
Drug: Bupivacaine
  Arms: Bupivacaine
Drug: liposomal bupivacaine
  Other Names: Exparel
  Arms: Liposomal bupivacaine

SUMMARY:
A prospective, randomized comparison of bupivacaine to liposomal bupivacaine given by local injection at all the wound sites in patients undergoing robotic-assisted or laparoscopic urologic surgeries in an effort to determine which method reduced postoperative opioid use the most.

DETAILED DESCRIPTION:
Liposomal bupivacaine was developed to extend the duration of efficacy of bupivacaine from the typical 6 - 8 hours up to 72 hours. The prolonged duration of liposomal bupivacaine was initially demonstrated in mice in 1994. Two randomized controlled trials using liposomal bupivacaine for bunionectomy and hemorrhoidectomy resulted in FDA approval for its use in humans. More recently, liposomal bupivacaine has also been found to improve pain control for patients undergoing total knee arthroplasty. Infiltration of a local anesthetic into laparoscopic port sites is a common practice that has been shown in some studies to improve postoperative pain. To compare liposomal bupivacaine and 0.25% bupivacaine for local analgesia following laparoscopic and robotic urologic surgery, a randomized comparison-controlled trial was performed.

ELIGIBILITY:
Inclusion Criteria:

* At least 18-years-old, undergoing laparoscopic urologic surgery.

Exclusion Criteria:

* Pregnant and/or nursing mothers.
* Allergy to bupivacaine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Knight, MD, Principal Investigator — San Antonio Uniformed Services Health Education Consortium
Locations (2):
- United States (2):
  - Baptist Health System, San Antonio, Texas
  - Methodist Healthcare System, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupivacaine: Surgical site infiltration of 0.25% bupivacaine.
  Bupivacaine
- Liposomal Bupivacaine: Surgical site infiltration of liposomal bupivacaine.
  liposomal bupivacaine
Period: Overall Study
Arm/Group | Bupivacaine | Liposomal Bupivacaine
Started | 100 | 106
Completed | 100 | 106
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Six patients were excluded from the 0.25% bupivacaine group: one for seizures; four for NSAID and/or PCA use; and one for incomplete data. Nine patients were excluded from the liposomal bupivacaine group; one for remaining intubated overnight; four for surgical complications; three for a hospital stay >5 days due to ileus; and one for NSAID use.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine | Liposomal Bupivacaine | Total
Number analyzed (Participants) | 94 | 97 | 191
Age, Customized [Median (Inter-Quartile Range); unit: years]
  Age | 63 [53 to 69] | 62 [52 to 68] | 63 [53 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 34 | 71
  Male | 57 | 63 | 120
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 45 | 55 | 100
  White | 41 | 32 | 73
  African American | 5 | 6 | 11
  Asian/Pacific Islander | 0 | 1 | 1
  Unknown | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 94 | 97 | 191
BMI [Median (Inter-Quartile Range); unit: kg/m2] | 28.9 [25.6 to 34.8] | 28.2 [25.5 to 32.8] | 28.7 [25.6 to 33.3]

OUTCOME MEASURES:

1. Primary Outcome: Total Opioid Consumption Measured in Intravenous Morphine Equivalents During the Postoperative Hospital Stay
Description: Total opioid consumption measured in intravenous morphine equivalents during the postoperative hospital stay
Time Frame: All data was recorded during the patient's hospital stay, typically less than 5 days. All data was tabulated from the electronic medical record, typically within 30 days of discharge from hospital.
Measure: Median (Inter-Quartile Range); unit: mg (morphine equivalents)
Arm/Group | Bupivacaine | Liposomal Bupivacaine
Number analyzed (Participants) | 94 | 97
mg (morphine equivalents) | 17.3 [8.3 to 30.5] | 15 [6.7 to 27]
Statistical Analysis 1: Comparison: Bupivacaine vs Liposomal Bupivacaine; Statistical analysis was performed using SAS, version 9.2 (Statistical Analysis Software, Cary, NC). All power calculations were at the 80% level with an alpha of 0.05. Based upon opioid consumption data previously reported for robotic-assisted laparoscopic prostatectomy, a sample size of 74 would be necessary to detect a 10 mg difference in morphine equivalents totaled over the entire hospital stay. (Webster TM, Herrell SD, Chang SS, et al. The Journal of Urology 2005;174(3):912-914; Test type: Superiority or Other; p = 0.39, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Visual Analog Pain Scores.
Description: Visual analog pain scores.
Time Frame: as for outcome 1
Reporting Status: Not Posted

3. Secondary Outcome: Length of Hospital Stay.
Description: Length of hospital stay.
Time Frame: as for outcome 1
Reporting Status: Not Posted

4. Secondary Outcome: Time to First Opioid Use.
Description: Time to first opioid use.
Time Frame: as for outcome 1
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Bupivacaine | Liposomal Bupivacaine
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/106
Other Adverse Events (participants affected / at risk) | 0/100 | 0/106

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No